CLINICAL TRIAL: NCT02965170
Title: Validation of a Laboratory Test Measuring Natalizumab (Tysabri®) Serum Levels in a Multiple Sclerosis Patient Cohort
Brief Title: Validation of a Laboratory Test Measuring Natalizumab (Tysabri®) Serum Levels in MS
Acronym: IIT12
Status: Completed | Type: Observational
Sponsor: Rocky Mountain MS Research Group, LLC (Other)
Collaborators: Abreos Biosciences (Other)
Responsible Party: Principal Investigator, John F. Foley, MD, Principal Investigator, Rocky Mountain MS Research Group, LLC
Other Study IDs: 001-012-TY
Record Dates: First submitted 2016-11-08; First posted 2016-11-16 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MS Tysabri: Patients with relapsing forms of multiple sclerosis and who are currently undergoing Tysabri® therapy at Rocky Mountain Multiple Sclerosis Research Group.

SUMMARY:
Validating a peptide-based laboratory test enabling the measurement of Tysabri® serum levels (pharmacokinetics, PK) in multiple sclerosis patients undergoing therapy. The results of this newly developed test will be compared to Tysabri® serum levels measured in parallel using an independent test. We will also simultaneously measure a pharmacodynamic marker of Tysabri®, receptor saturation levels on blood immune cells, which is thought to correlate with Tysabri® serum levels.

DETAILED DESCRIPTION:
From a single site, consenting patients with relapsing forms of multiple sclerosis who are currently begin treated with Tysabri® (natalizumab) and meeting the eligibility criteria will be asked to provide blood samples on the same day, and prior to, a scheduled infusion of Tysabri® 300 mg IV. Up to 500 patients will be enrolled in this study. Each patient may be asked to donate blood up to 2 times (one blood draw per cycle) to obtain longitudinal data points. Each patient will also be asked to fill out a wellness patient reported outcome (PRO) questionnaire along with the blood draws

ELIGIBILITY:
Inclusion Criteria:

* Infusing with Tysabri at a single site, Rocky Mountain MS Clinic

Exclusion Criteria:

* If subject donated or received blood, plasma, or any other blood products between the last Tysabri® infusion and the time of sample collection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients with multiple sclerosis who have had one or more doses of Tysabri® (natalizumab) and are currently being treated with Tysabri® will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Natalizumab Concentrations in Serum | 12 Months
  Validate a novel peptide-based laboratory test enabling the measurement of nadir natalizumab (Tysabri®) serum levels in multiple sclerosis patients undergoing therapy compared to the traditional ELISA assay

CONTACTS AND LOCATIONS:
Overall Officials: John F Foley, MD, Principal Investigator — Rocky Mountain MS Research Group
Locations (1):
- Rocky Mountain MS Clinic, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No